CLINICAL TRIAL: NCT05593926
Title: Fibre suppLements fOR Pre-diAbetes
Brief Title: Fibre suppLements fOR Pre-diAbetes - An Assessment Oral Fibre Supplements on Pre-diabetes Outcome Measures
Acronym: FLORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Myota GmbH (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Principal Investigator, Dr John Luke Twelves, Medical Director (CRO), Myota GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LH005
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Two-arm, individually randomized, single-blind placebo-controlled trial
Who Masked: Participant
Masking Description: Participants will be randomised to Placebo or the Myota Metabolic Regulator, with a 1:1 randomisation ratio stratified by gender and BMI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The functional food, Myota Metabolic Regulator, consisting of 20g of a powdered fibre mix, to be taken daily alongside usual diet for 24 weeks.
  Interventions: Dietary Supplement: Myota Metabolic Regulator
- Placebo (No Intervention): Placebo will be 2g of powdered cellulose, to be taken daily alongside usual diet for 24 weeks. Placebo will be 2g of powdered cellulose, to be taken daily alongside usual diet for 24 weeks.

INTERVENTIONS:
Dietary Supplement: Myota Metabolic Regulator — The functional food, Myota Metabolic Regulator, consisting of 20g of a powdered fibre mix, to be taken daily alongside usual diet for 24 weeks.
  Arms: Intervention

SUMMARY:
This trial will investigate whether a powdered fibre mix helps maintain healthy blood glucose levels in participants with pre-diabetes, where high blood sugar is a risk of diabetes.

DETAILED DESCRIPTION:
Pre-diabetes is characterised by high blood glucose levels, high plasma cholesterol, low-density lipoprotein (LDL) and high-density lipoprotein (HDL). Dietary fibre consumption has been hypothesised to improve these metabolic parameters through the viscous properties, and the production of short-chain fatty acids (SCFA) in the intestine.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Have a Body Mass Index (BMI) of at least 25 kg/m2
* Men or post menopausal* women aged 18-70
* Identified as pre-diabetic (HbA1c 6.0% (42 mmol/mol) to 6.4% (47 mmol/ mol)) within the previous 12 months
* Baseline HbA1c result within the range 5.8% (40 mmol/mol) - 6.5% (48 mmol/mol)
* Willing to complete in clinic blood tests and a participant trial survey
* Have access to a smartphone or a computer

Exclusion Criteria:

* Receiving medication to treat Type 1 or Type 2 diabetes in the previous 6 months
* Have a Body Mass Index (BMI) <25 kg/m2 and >45 kg/m2
* Loss of more than 5% body weight in last 3 months
* Current participation in weight loss program or planned in the next 16 weeks
* Steroid use (except for over the counter NSAID's, topical steroids and inhalers)
* Severe hepatic diseases (including chronic persistent hepatitis, liver cirrhosis or the co-occurrence of positive hepatitis B virus surface antigen and abnormal hepatic transaminase (serum concentrations of alanine transaminase or aspartate transaminase >2.5× the upper normal limit))
* Continuous antibiotic use for >3 days within 4 weeks prior to enrolment
* Continuous use of weight-loss drug for within 3 months of study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
HbA1c levels | 16 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on Hemoglobin A1c (HbA1c) levels

SECONDARY OUTCOMES:
HbA1c levels | 24 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on Hemoglobin A1c (HbA1c) levels
Insulin | 16 and 24 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on blood insulin concentration.
Insulin sensitivity | 16 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on insulin sensitivity as measured using ISI-OGTT.
Lipid profile | 16 and 24 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on cholesterol [total, low-density lipoprotein (LDL), high-density lipoprotein (HDL)] and triglycerides levels.
Inflammatory markers | 16 and 24 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on inflammatory markers (IL-6, IL-8, IL-10, CRP, TNF-a).
Blood pressure | 16 and 24 weeks
  To compare the effect of Myota's Metabolic Regulator versus placebo on diastolic and systolic blood pressure
Overall safety of the Myota Metabolic Regulator | Weeks 1-4
  Number of participants reporting adverse events (AEs) and serious adverse events (SAEs)
To investigate intervention adherence | 24 weeks
  A daily intervention adherence questionnaire will be used to assess the extent to which participant's adhered to the intervention. This will consist of two questions:
  Did you consume the full sachet of study product yesterday? Yes/No [If no] Why were you unable to take the product yesterday?
To investigate usability | 16 and 24 weeks
  A usability questionnaire will be administered to assess how easily participant's were able to use the intervention or placebo. This will consist of two statements:
  I found the supplement easy to take. Strongly disagree to Strongly agree (5 options) I would like to take this supplement in my normal daily life. Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Luke Twelves, Dr, Principal Investigator — Myota GmbH; Thomas Gurry, PhD, Study Director — Myota GmbH
Locations (2):
- United Kingdom (2):
  - Albany House Medical Centre, Wellingborough, Northamptonshire
  - Lindus Health, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall CV, Twelves JL, Saxena M, Scapozza L, Gurry T. Effects of a diverse prebiotic fibre supplement on HbA1c, insulin sensitivity and inflammatory biomarkers in pre-diabetes: a pilot placebo-controlled randomised clinical trial. Br J Nutr. 2024 Jul 14;132(1):68-76. doi: 10.1017/S0007114524000904. Epub 2024 Apr 24. PMID 38654680

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT05593926/SAP_002.pdf